CLINICAL TRIAL: NCT02411227
Title: Evaluation of Neurocognitive Driving Rehabilitation in Virtual Environments (NeuroDRIVE) as an Adjunctive Intervention for Traumatic Brain Injury
Brief Title: Neurocognitive Driving Rehabilitation in Virtual Environments (NeuroDRIVE) as an Adjunctive Intervention for Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: The Center for Neuroscience and Regenerative Medicine (CNRM) (Unknown); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150103; 15-CC-0103
Record Dates: First submitted 2015-04-07; First posted 2015-04-08 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Traumatic Brain Injury
Keywords: Neuropsychologic Testing; Neurocognitive; Virtual Reality; Rehabilitation; Driving
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Immediate Intervention
  Interventions: Behavioral: VR Driving
- 2 (No Intervention): Wait list

INTERVENTIONS:
Behavioral: VR Driving — Baseline: Tactical A3 scenario, composite score Post-Assessment: Tactical A4 scenario composite score
  Arms: 1

SUMMARY:
Background:

- People with traumatic brain injury (TBI) can have problems with thinking and everyday activities. They may have a higher risk for car accidents. NeuroDRIVE uses a virtual reality driving simulator. Researchers think it can help test and improve how people think and drive after TBI.

Objective:

- To test how NeuroDRIVE affects brain performance and driving safety.

Eligibility:

- People at least 18 years old with a history of TBI and who had a driver s license at some point. They must speak, read, and write English and be physically able to drive.

Design:

* Participants will be asked to release their driving records, but they do not have to do this to be in the study.
* Visit 1: Screening physical exam.
* Visit 2: Magnetic resonance imaging (MRI) scan. Participants will lie on a table that slides into a cylinder with a strong magnetic field. A device will be placed over the head. Participants may do computer tasks during the scan.
* Participants will have tests of memory, attention, and thinking. They may be asked questions, take tests, and do simple actions.
* Visit 3: Tests of memory, attention, and thinking, plus a virtual reality driving assessment.
* Participants will be assigned to Group 1 to start NeuroDRIVE training immediately or Group 2 to start 10 weeks later.
* Visits 4 9, over 4 weeks:
* Participants will practice driving skills and mental exercises in the simulator.
* They will complete a driving questionnaire online each week.
* Visit 10: Repeat of Visit 3, with some small changes.
* Visits 11-12: Very similar to Visits 1-2. Includes MRI scan; physical exam; questionnaires; and tests of thinking, memory, and attention..
* After Visit 12: Participants will fill out a weekly driving survey online for 4 weeks.

DETAILED DESCRIPTION:
OBJECTIVE:

The primary objective of this study is to evaluate the NeuroDRIVE behavioral intervention for enhancement of driving abilities, cognitive abilities, and neurobehavioral symptoms after traumatic brain injury (TBI). For the purposes of this protocol, NeuroDRIVE refers to the novel combined approach of driving training and cognitive rehabilitation in a virtual reality environment. While NeuroDRIVE utilizes the VR system as the method through which the intervention is administered, NeuroDRIVE is not the VR system itself.

STUDY POPULATION:

30 adult patients with a history of mild TBI and 30 adult patients with a history of moderate-to-severe TBI. Participants will be recruited from the National Institutes of Health (NIH), WRNMMC, and the broader community.

DESIGN:

The current study is a Clinical Trial Phase II interventional research study. The primary purpose of the study is for treatment, and it will employ a parallel intervention model. There will be no masking (i.e., open label). Participants will be classified into two groups by TBI severity: those with history of mild TBI and those with history of moderate-tosevere TBI. These different severities are known to have distinct cognitive sequelae. Within each severity group, participants will be in a 2 (pre-post) x 2 (treatment vs. wait list) experimental design.

OUTCOME MEASURES:

Primary outcome measures will include:

* Results from the Virtual Reality Driving Assessment (baseline and postintervention Tactical scenario composite scores)
* Total scores on the Neurobehavioral Symptom Inventory
* Standard and scaled scores from the following cognitive assessments (from the TBI Common Data Elements identified by NINDS):

WAIS-IV or WMS-IV Digit Span subtest

WAIS-IV Digit-Symbol Coding subtest

Secondary outcome measures will include:

-Neuroimaging results:

Regions of Interest for FMRI: Bilateral dorsolateral prefrontal cortex

Regions of Interest for DTI: Corpus callosum, bilateral frontal white matter horns, and bilateral longitudinal fasciculi

-Total scores on the following symptom questionnaires:

Glasgow Outcome Scale-Extended (GOS-E)

Ohio State University TBI Identification Method

Brief Symptom Inventory- 18

Satisfaction with Life Scale (SWLS)

PTSD Checklist- Civilian (PCL-C)

SF-36v2 Health Survey (SF-36v2)

Fatigue Severity Scale (FSS)

Epworth Sleepiness Scale (ESS)

Beck Depression Inventory-II (BDI-II)

Combat Exposure Scale (CES)

Dual Dangerous Driving Index (DDDI)

-Standard and scaled scores from the following cognitive phenotyping assessments (from the TBI Common Data Elements identified by NINDS):

California Verbal Learning Test- Second Edition (CVLT-II)

WAIS-IV Symbol Search subtest

Medical Symptom Validity Test (MSVT)

-Standard and scaled scores from the following additional cognitive phenotyping assessments:

Trail Making Test (TMT)

Test of Premorbid Functioning (ToPF)

Grooved Pegboard

Controlled Oral Word Association Test (COWAT)

Bethesda Eye and Attention Measure (BEAM)

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects eligible for participation must meet the following criteria:

1. Currently has a valid driver s license, or had a valid driver s license prior to injury
2. 18 years of age or older
3. Able to effectively manipulate the steering wheel and the gas/brake pedals without adaptive equipment
4. Able to read, write, and speak in English
5. History of traumatic brain injury greater than 12 weeks prior to initiation into the current study
6. Able to provide informed consent
7. NBSI score greater than or equal to 16 (Mild TBI sub-group only)

EXCLUSION CRITERIA:

Subjects are not eligible for participation if any of the following conditions exist:

1. Risk for injury from the MRI magnet, including:

   * Pacemakers or other implanted electrical devices.
   * Brain stimulators.
   * Some types of dental implants.
   * Aneurysm clips (metal clips on the wall of a large artery).
   * Metallic prostheses (including metal pins and rods, heart valves, and cochlear implants).
   * Permanent eyeliner (other non-metallic tattoos are permissible).
   * Implanted delivery pump.
   * Shrapnel fragments.
   * Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye of which they may be unaware.
   * Fear of confined spaces.
   * Back problems that may result in back pain or discomfort from lying in the scanner.
   * Weight of over 350 pounds, due to the weight limit of the MRI table.
   * It is not known if MRI is completely safe for a developing fetus. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each MRI scan. The scan will not be done if the pregnancy test is positive. Because neuroimaging is a key component of the current study, inability to participate in MRI scanning is a necessary exclusion criterion.
2. History of penetrating brain injury
3. History of serious medical condition other than TBI that could affect cognitive or motor abilities (e.g., multiple sclerosis, encephalitis, cerebrovascular disease)
4. History of severe motion sickness and/or vertigo.
5. Other medical or psychological instability that could create difficulty fulfilling the study requirements (e.g., untreated mental illness, auditory/visual hallucinations, narcolepsy)

To verify this information, study coordinators will request medical records (i.e., recent medical history, medication list, any neuroimaging, and records pertinent to the participant s recent injury) to further evaluate potential participants inclusion into the study. Medical records can be obtained in three ways:

1. Participants can bring the records when they come to NIH for testing; it will be made clear if they do not bring this information with them and we cannot verify that they meet inclusion criteria, potential participants will not be enrolled into the study that day.
2. Alternatively, the participants can also fax their medical records to a secured fax machine at the Recreational Therapy office at the NIH where access is only permitted to study staff (i.e., scheduler, physician, and nurse psychologist).
3. Participants may also fill out a medical release document and submit it to the study coordinator.

Medical history data will be reviewed, and if it is clear that the patient does not meet the inclusion criteria, we will contact them and cancel their appointment. Data obtained in this manner may be used to evaluate participant eligibility; however, it will not be used for any research purposes. Additionally, for any patients who are deemed not eligible to participate, their medical history data will be destroyed in accordance with NIH regulations.

As a condition of receiving funding from CNRM, de-identified imaging and phenotyping data (i.e., neurocognitive test results and behavioral questionnaires) from funded studies must be made available within a centralized repository (the CNRM Informatics Core) one year after the completion of the study. This is intended to facilitate use and analysis of this data for future research questions or projects. As such, potential subjects will be informed that they should not participate in this study if they do not want their data used for other projects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
VR Driving, Cognitive test, and Symptoms | pre/post after 16 weeks of intervention
  -Results from the Virtual Reality Driving Assessment (baseline and post- intervention Tactical scenario composite scores)-Total scores on the Neurobehavioral Symptom Inventory-Standard and scaled scores from the following cognitive assessments (from the TBI Common Data Elements identified by NINDS):--WAIS-IV Digit Span subtest--WAIS-IV Digit-Symbol--Coding subtest

SECONDARY OUTCOMES:
MRI, Phenotyping, & Driving evals | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Leighton Chan, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ortoleva C, Brugger C, Van der Linden M, Walder B. Prediction of driving capacity after traumatic brain injury: a systematic review. J Head Trauma Rehabil. 2012 Jul-Aug;27(4):302-13. doi: 10.1097/HTR.0b013e3182236299. PMID 21897289
- [Background] Cox DJ, Davis M, Singh H, Barbour B, Nidiffer FD, Trudel T, Mourant R, Moncrief R. Driving rehabilitation for military personnel recovering from traumatic brain injury using virtual reality driving simulation: a feasibility study. Mil Med. 2010 Jun;175(6):411-6. doi: 10.7205/milmed-d-09-00081. PMID 20572473
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-CC-0103.html